CLINICAL TRIAL: NCT06726044
Title: Effectiveness of Rehabilitation After Arthroscopic ACL Reconstruction Using Inertial Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University in Zielona Góra (Other)
Collaborators: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Mariusz Naczk, Professor, University in Zielona Góra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: University of Zielona Gora
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: ACL reconstruction
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: The study finally included 24 people after ACL reconstruction. All of them participated in 12 - week rehabilitation; SR - standard rehabilitation, SR+I - standard rehabilitation and inertial exercises
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard rehabilitation (Active Comparator): 12 subjects after ACL reconstruction. Subjects participated in standard rehabilitation program twice a week for 12 weeks. Each session lasted approximately 60 minutes.
  Interventions: Other: Standard rehabilitaion after ACL reconstruction; Other: Standard rehabilitaion after ACL reconstruction plus inertial exercises
- Standard rehabilitation and inertial exercises (Experimental): 12 subjects after ACL reconstruction. Subjects participated in standard rehabilitation program twice a week for 12 weeks and additionally performed inertial exercises from the fifth week of rehabilitation. Then each session lasted approximately 70 minutes.
  Interventions: Other: Standard rehabilitaion after ACL reconstruction; Other: Standard rehabilitaion after ACL reconstruction plus inertial exercises

INTERVENTIONS:
Other: Standard rehabilitaion after ACL reconstruction — The SR group, consisting of 12 participants, underwent a standard rehabilitation program twice a week for 12 weeks. Each session lasted approximately 60 minutes and was conducted by the same therapist.
  After 12 weeks of rehabilitation, effectiveness was evaluated using standard tests. Before rehabilitation involving kinesiotherapy (two weeks post-surgery), the following measurements were conducted:
  Height and body weight Thigh circumference measurements Assessment of muscle and tendon stiffness Body composition evaluation
  After the rehabilitation the following measurements and assessments were conducted:
  Body weight Thigh circumference measurements Assessment of muscle and tendon stiffness Body composition evaluation Evaluation of the strength of knee extensor and flexor muscles under isokinetic conditions Evaluation of knee extensor strength under inertial conditions Postural stability assessment
Other: Standard rehabilitaion after ACL reconstruction plus inertial exercises — The SR+I group, consisting of 12 participants, underwent a standard rehabilitation program twice a week for 12 weeks including inertial exercises. Each session lasted approximately 70 minutes and was conducted by the same therapist.
  Subjects also performed inertial exercises from the fifth week of rehabilitation. These exercises were conducted on an InerKnee. The inertial exercises protocol included: knee extension exercises performed in a seated position for the operated leg, 4 sets of exercises, each lasting 15 seconds individually, adjusted resistance to maintain a 1-second extension cycle, passive rest periods of 2 minutes between sets After 12 weeks of rehabilitation, effectiveness was evaluated using standard tests the same as in SR group.

SUMMARY:
The primary aim of the study was to compare the effectiveness of two rehabilitation protocols for patients following ACL reconstruction. The first group (SR) underwent standard rehabilitation, which included the following treatments:

Manual therapy: manual mobilization of the patella and fibular head Anti-swelling therapy: manual lymphatic drainage techniques Compression and cryotherapy Reflex therapy: clavi-therapy Kinesiotherapy: strength exercises Kinesiotaping Osteopathic techniques Myofascial release Manual scar treatment Activation of gliding movement in the knee joint; soft tissue techniques in the popliteal region Flossing Knee flexion and extension exercises in a closed and next in open kinematic chain Isometric quadriceps exercises at full extension and 45-degree flexion

In addition to the above, the second group (SR+I) performed inertial exercises, which were introduced starting from the fifth week of rehabilitation. After 12 weeks of rehabilitation, its effectiveness was evaluated using standard tests.

The results indicate that the innovative rehabilitation protocol incorporating inertial exercises can be effectively applied in the rehabilitation of individuals following arthroscopic ACL reconstruction. None of the monitored rehabilitation effectiveness indicators in the SR+I group were inferior to those in the SR group. Moreover, certain parameters assessing rehabilitation effectiveness showed the SR+I protocol to have advantages over the SR protocol.

DETAILED DESCRIPTION:
The primary goal of the study was to compare the effectiveness of two rehabilitation protocols in patients following ACL reconstruction. The first group (SR), consisting of 12 participants, underwent a standard rehabilitation program twice a week for 12 weeks. Each session lasted approximately 60 minutes and was conducted by the same therapist. The standard rehabilitation program included the following treatments:

Manual therapy: manual mobilization of the patella and fibular head Anti-swelling therapy: manual lymphatic drainage techniques Compression and cryotherapy Reflex therapy: clavi-therapy Kinesiotherapy: strength exercises Kinesiotaping Osteopathic techniques Myofascial release Manual scar treatment Activation of gliding movement in the knee joint; soft tissue techniques in the popliteal region Flossing Knee flexion and extension exercises in closed kinematic chains The same in open kinematic chains Isometric quadriceps exercises at full extension and 45-degree flexion

The second group (SR+I) followed the same standard protocol but also performed inertial exercises from the fifth week of rehabilitation. These exercises were conducted on an InerKnee setup, adapted from the Cyklotren device, and began four weeks post-surgery, provided the patient achieved at least 90 degrees of knee flexion (including full extension). The inertial exercises protocol included:

knee extension exercises performed in a seated position for the operated leg 4 sets of exercises, each lasting 15 seconds individually adjusted resistance to maintain a 1-second extension cycle passive rest periods of 2 minutes between sets

After 12 weeks of rehabilitation, effectiveness was evaluated using standard tests. The results showed that the innovative rehabilitation protocol, incorporating inertial exercises, can be effectively applied to patients following arthroscopic ACL reconstruction. No monitored indicators in the SR+I group were worse than those in the SR group. In fact, several parameters indicated the SR+I protocol's superiority over the standard protocol.

ELIGIBILITY:
Inclusion Criteria:

* ACL reconstruction performed by the same doctor using similar technique, lack of other disases, minimum 90% attendance in rehabilitation sessions

Exclusion Criteria:

* other chronic disases, rehabilitation was not completed, other injury during rehabilitation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-04-02 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Knee extensors anf flexors strength under isokinetic and inertial conditions. | 12 weeks of rehabilitation
  After 12 weeks of rehabilitation, muscle strength was assessed in all patients under isokinetic and inertial conditions. Measurements were conducted following these guidelines:
  * Isokinetic measurements at two speeds: of 60˚/s, and 180˚/s, with five repetitions of flexion and extension for each limb and each speed in a seated position,
  * the axis of rotation of the dynamometer was aligned with the axis of rotation of the knee joint.
  * patients performed trial repetitions to familiarize themselves with the movement speed and range of motion.
  the range of motion was consistently set at 60˚, starting from a knee flexion angle of 90˚ ± 30˚.
  * patients were secured using crossed straps, a hip belt, and a limb-specific belt.
  * only the patient and the examiner are allowed in the room during the measurement process
  The patient's arms were crossed on the chest during the measurement. Testing began with the healthy limb and concluded with the operated limb. Patients

SECONDARY OUTCOMES:
Body balance, stability and mobility after rehabilitation | 12 weeks of rehabilitation
  Y-Balance Test - Examination Description
  The Y-Balance Test is a dynamic balance assessment tool used to evaluate an individual's postural control and stability. Here's the procedure:
  * positioning: the participant stands on a designated mark with one foot (the tested limb), which serves as the base and starting point for all three arms of the Y-shape scale. The opposite foot (non-tested limb) is used to reach as far as possible along the measurement arms of the Y.
  * testing directions: Anterior Posterolateral Posteromedial
  * rules: the foot of the reaching limb must not bear weight or touch the floor forcefully. The arms must stay positioned on the hips during the entire test. Loss of balance, ground contact with the reaching foot, or incorrect arm positioning invalidates the trial
  * execution: the participant performs three attempts for each direction. The farthest distance reached in each direction is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Education and Sport, Faculty in Gorzow Wielkopolski, Poznan University of Physical Education, Poznan, Poland, Gorzów Wielkopolski, Poland

IPD SHARING:
Plan to Share IPD: Yes
All data from research excluding private data; names etc.
Supporting Information: Study Protocol, CSR
Time Frame: After publication these data in article, we suppose from 2025
Access Criteria: from the corresponding author